CLINICAL TRIAL: NCT05556993
Title: Parkinson's Research With Inclusion, Diversity and Equity
Acronym: PRIDE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Sponsor
Other Study IDs: UNLV-2021-265
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Caregiver; Health care provider; LGBTQIA+
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- LGBTQIA+ Persons living with Parkinson's Disease: 125 LGBTQIA+ persons living with Parkinson's Disease will be asked to do a 45-minute phone survey.
- Non- LGBTQIA+ Persons living with Parkinson's Disease: 125 Non- LGBTQIA+ persons living with Parkinson's Disease will be asked to do a 45- minute phone survey.
- LGBTQIA+ caregivers of people living with Parkinson's Disease: 125 LGBTQIA+ caregivers of people living with Parkinson's Disease will do a 45-minute phone survey.
- Non- LGBTQIA+ caregivers of people living with Parkinson's Disease: 125 non- LGBTQIA+ caregivers of people living with Parkinson's Disease will do a 45-minute phone survey.
- Health care providers of people living with Parkinson's Disease: 100 health care providers of people living with Parkinson's Disease will complete a 45-minute online survey.

SUMMARY:
The purpose of this study is to identify the health and healthcare needs of LGBTQIA+ and non LGBTQIA+ communities living with Parkinson's disease.

DETAILED DESCRIPTION:
Four million LGBTQIA+ adults age 50+ live in the U.S. Very little is known about the needs of the LGBTQIA+ community living with Parkinson's disease (PD). This research will work with the LGBTQIA+ community to learn about the health needs of those living with PD. The researchers will also talk to caregivers about their care experiences, and ask healthcare providers about their work with LGBTQIA+ communities living with PD. LGBTQIA+ adults have more health and care problems. This study will test if LGBTQIA+ adults with PD experience more health and care problems. This study will also see if caregivers have more problems and how providers are caring for the LGBTQIA+ community living with PD. LGBTQIA+ adults living with PD, caregivers and care providers will be asked to fill out a survey. Some caregivers will be asked to participate in an hour interview to learn about their experiences. Surveys and interviews can be done by phone or internet. The study will find ways to improve health and care of LGBTQIA+ people living with PD. The study will share findings so others can help to make care better for the LGBTQIA+ community.

ELIGIBILITY:
Inclusion Criteria:

* Identify as LGBTQIA+ or non-LGBTQIA+
* Aged 18+
* Ability to complete the phone or online survey in English/Spanish
* Diagnosis of Parkinson's disease or a caregiver of a person with Parkinson's disease
* Health care professional that provides care to patients living with Parkinson's disease

Exclusion Criteria:

* Not having a diagnosis of Parkinson's disease
* Not currently or in the past a caregiver of a person with Parkinson's disease
* Not currently providing care to patients with Parkinson's disease
* Inability to complete the survey in English or Spanish
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population includes individuals aged 18 and older who identify as lesbian, gay, bisexual, transgender, queer, intersex and/or another identity (LGBTQIA+) and non-LGBTQIA+ persons living with Parkinson's disease and their caregivers, as well as health care professional, including physicians, physician assistants, nurse practitioners, psychologists, physical or occupational therapists, registered nurses, social workers, and others, who provide care to persons living with Parkinson's disease.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-06-29 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Depressive Symptoms | Baseline
  Depressive symptoms will be measured by Patient Health Questionnaire nine items, with higher scores indicating a higher frequency of depressive symptoms
Parkinson's Disease Symptoms | Baseline
  Severity of Parkinson's Disease will be measured by Movement Disorder Society Unified Parkinson's Disease Rating Scale Parts one and two, with higher scores suggesting more severe Parkinson's disease symptoms
Health-related quality of life | Baseline
  Quality of Life is measured by Parkinson's Disease Quality of Life Questionnaire Summary Index eight items, with higher scores indicating worse quality of life
Cognition | Baseline
  Cognition is measured by Telephone Interview for Cognitive Status nine items, with lower scores indicating potential cognitive impairment
Caregiver Burden | Baseline
  Caregiver Burden is measured by Zarit Caregiver Burden Inventory twelve items, with higher scores representing more burden
Cultural Competency of Health Care Providers | Baseline
  Cultural competency is measured by Lesbian, Gay, Bisexual, Transgender Development of Clinical Skills Scale eighteen items, with higher scores indicating higher levels of clinical preparedness and less prejudicial attitudinal awareness regarding LGBT patients

CONTACTS AND LOCATIONS:
Overall Officials: Jason Flatt, PhD, Principal Investigator — University of Nevada, Las Vegas
Locations (1):
- University of Nevada, Las Vegas, Las Vegas, Nevada, United States

REFERENCES:
- [Background] Lin CR, Rosendale N, Deeb W. Expanding sexual and gender minority research in movement disorders: More than awareness and acceptance. Parkinsonism Relat Disord. 2021 Jun;87:162-165. doi: 10.1016/j.parkreldis.2021.05.019. Epub 2021 May 24. PMID 34088617
- [Background] Rosendale N, Wong JO, Flatt JD, Whitaker E. Sexual and Gender Minority Health in Neurology: A Scoping Review. JAMA Neurol. 2021 Jun 1;78(6):747-754. doi: 10.1001/jamaneurol.2020.5536. PMID 33616625
- [Background] Anderson JG, Flatt JD. Characteristics of LGBT caregivers of older adults: Results from the national Caregiving in the US 2015 survey. Journal of Gay & Lesbian Social Services. 2018;30(2):103-116.